CLINICAL TRIAL: NCT06657365
Title: Safety and Efficacy Evaluation of the Monopolar Radiofrequency Device for the Improvement of the Facial Wrinkles, a Prospective, Multicenter, Evaluator Blinded, Randomized, Parallel-controlled, Non-inferior Clinical Trial
Brief Title: Safety and Efficacy Evaluation of the Monopolar Radiofrequency Device for the Improvement of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CLASSYS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLSSPZLY
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Facial Wrinkles; Anti-Aging; Wrinkles and Rhytides; Wrinkles Such as Nasolabial Folds; Wrinkles
Keywords: VOLNEWMER; facial skin treatment; nasolabial folds; marionette line; MRF; facial wrinkles; wrinkles; monopolar radiofrequency device
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VOLNEWMER (Experimental): A non-invasive skin tightening treatment using the Volnewmer device.
  Interventions: Device: Radiofrequency (RF) Treatment with Volnewmer
- Thermage CPT (Active Comparator): A non-invasive skin tightening treatment using the Thermage CPT device.
  Interventions: Device: Radiofrequency (RF) Treatment with Thermage CPT

INTERVENTIONS:
Device: Radiofrequency (RF) Treatment with Volnewmer — Non-invasive radiofrequency-based skin tightening using the Volnewmer device.
  Arms: VOLNEWMER
Device: Radiofrequency (RF) Treatment with Thermage CPT — Non-invasive radiofrequency-based skin tightening using the Thermage CPT device.
  Arms: Thermage CPT

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of the monopolar radiofrequency therapy device developed by CLASSYS Inc. for improving facial and periorbital wrinkles. This is a prospective, multicenter, evaluator-blinded, randomized, parallel-controlled, non-inferiority clinical trial.

The main questions the study aims to answer are:

Does the monopolar radiofrequency device improve the appearance of facial and periorbital wrinkles? Is the safety profile of the monopolar radiofrequency device acceptable?

Researchers will compare the investigational device to the Thermage CPT System (Solta Medical Co., Ltd.) to see if the monopolar radiofrequency device is non-inferior in terms of wrinkle improvement.

Participants will:

Undergo a single treatment session with either the investigational device or the control device.

Be followed up for a period of 3 months to assess wrinkle improvement and safety outcomes.

The primary outcome will be the improvement in facial and periorbital wrinkles, measured by the Facial Wrinkle and Elasticity Scale (FWES), 3 months post-treatment. Secondary outcomes include the Global Aesthetic Improvement Scale (GAIS) and a Visual Analog Scale (VAS) for pain. Safety evaluations will include adverse event (AE) and serious adverse event (SAE) monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old（The date of signing the informed consent shall prevail）, gender is not limited.
2. Facial and periorbital wrinkle and elasticity Scale (FWES) Score ≥ 3 points. Both the facial and periorbital FWES should meet the criteria.
3. The subject fully understands the benefits and risks of this experiment, and is still willing to participate and sign the informed consent.

Exclusion Criteria:

1. Individuals with skin diseases, scars, open wounds, or metal implants in the area where clinical trial medical devices will be applied.
2. Patients with implanted electrical devices (e.g., pacemakers, AICDs).
3. Those with a history of hypertrophic scars, keloids, or severe allergic reactions.
4. Individuals with excessive facial fat requiring surgical treatment.
5. Those with autoimmune diseases, acute viral herpes, or poorly controlled diabetes.
6. People with abnormal coagulation function or those taking anticoagulant medications (e.g., aspirin, warfarin) within 1 week of screening.
7. Individuals treated with fillers or botulinum toxin within the last 6 months or permanent fillers in the treatment area.
8. Those who have received skin treatments (e.g., deep exfoliation, lasers, light therapy) in the treatment area within 6 months.
9. Pregnant or lactating women, or women of childbearing potential not using medically accepted contraception.
10. Persons deemed inappropriate by the investigator to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
FWES | 3 months after the treatment
  Facial wrinkle improvement was defined as reduction of FWES subgroup score≥1.

CONTACTS AND LOCATIONS:
Overall Officials: 文志 李, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital[北京安贞医院], Beijing, China